CLINICAL TRIAL: NCT01123759
Title: Consuming Fish to Reduce Mercury Intake While Optimizing Omega-3 Fatty Acid Status
Brief Title: Healthful Seafood Consumption for Sensitive Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Florida A&M University (Other)
Responsible Party: Charles Santerre, Professor, Purdue University, Dept of Foods and Nutrition
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USDA-CSREES 07-5110-03804
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Infant Brain Health
Keywords: Fish; mercury; omega-3 fatty acids; infant; brain development; pregnancy; nursing mother; dietary recommendations; Hair mercury; Blood mercury; Recommendations for pregnant or nursing women; Infant brain health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tilapia (Active Comparator): Subjects are fed 6 oz tilapia once a week for 3 months
  Interventions: Other: Feeding low mercury fish
- Salmon (Active Comparator): Subjects fed 6 oz salmon once a week for 3 months
  Interventions: Other: Feeding low mercury fish

INTERVENTIONS:
Other: Feeding low mercury fish — Subjects fed 6 oz of either tilapia (low omega-3 fish) or salmon (high omega-3 fish) for 3 months. Both fish are low in mercury

SUMMARY:
Fish can provide pregnant women with omega-3 fatty acids for fetal brain development but some fish contains high levels of mercury which is detrimental to fetal brain development. The hypothesis is that women who have previously consumed high mercury fish can reduce the mercury level in their bodies and improve their omega-3 levels in three months by eating fish that is high in omega-3 fatty acids and low in mercury.

DETAILED DESCRIPTION:
Exposure to methylmercury, a developmental toxicant found primarily in fish. Fish is nutritionally important for providing long chain omega-3 fatty acids that are important for perinatal health. Since maternal transfer of mercury and omega-3 fatty acids are the primary routes for fetal (placental transfer) or infant (maternal milk) exposure, there is a critical need to develop specific advice for childbearing-aged women based upon the 2004 Dietary Guidelines Advisory Committee's recommended intake i.e., consume 8 ounces of fish per week. This clinical trial investigates whether weekly consumption of selected fish species for 12 weeks can improve plasma concentrations of the omega-3 fatty acids (eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA)) while reducing hair or blood mercury concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Hair mercury levels equal to or greater than 0.8 ppm

Exclusion Criteria:

* Pregnant or planning to become pregnant in the next 3 months
* Nursing

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Hair Mercury | 3 months
  The hair mercury after feeding low mercury fish for 3 months

SECONDARY OUTCOMES:
Blood mercury concentration | 3 months
  The blood mercury concentration after feeding low mercury fish for 3 months
Blood omega-3 fatty acid concentrations | 3 months
  Blood omega-3 fatty acid concentration after feeding either salmon or tilapia for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles Santerre, Ph.D, Principal Investigator — Purdue University, Department of Foods and Nutrition
Locations (2):
- United States (2):
  - Florida A&M University, Tallahassee, Florida
  - Purdue University, Department of Foods and Nutrition, West Lafayette, Indiana